CLINICAL TRIAL: NCT01411410
Title: A Phase 1 Study of BAY80-6946 (Phosphatidylinositol 3΄-Kinase Inhibitor) in Combination With Paclitaxel in Subjects With Advanced Solid Malignancy
Brief Title: Phase I Study of PI3(Phosphoinositol 3)-Kinase Inhibitor BAY80-6946 With Paclitaxel in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12874
Record Dates: First submitted 2011-08-05; First posted 2011-08-08 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Neoplasms
Keywords: phase I; phosphatidylinositol 3΄-kinase (PI3K); paclitaxel; Maximum tolerated Dose
MeSH Terms: conditions — Neoplasms | interventions — Paclitaxel; copanlisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Copanlisib (BAY80-6946) (Experimental): The treatment of consists of repetitive cycles, each over 4 weeks. It continues until disease progression or limiting toxicity. If paclitaxel is discontinued for toxicity, BAY80-6946 may continue at the discretion of the investigator if a clinical benefit (response or stable disease for 6 months) is noted.
  Interventions: Drug: Paclitaxel; Drug: Copanlisib (BAY80-6946)

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel (80 mg/m2 in Cohort 1, 2 and 3, 90 mg/m2 in Cohort 4) as 60-minute iv infusion once weekly on Days 1, 8, 15 and 22 (Day 22 in Cohort 1, 2 and 3 only) in 28-day cycles
  * The following intravenous premedications are required 30 to 60 minutes before paclitaxel infusion: Dexamethasone (10 mg), diphenhydramine (50 mg) and either cimetidine (300 mg) or ranitidine (50 mg)
  * Alternatively, for premedications other than dexamethasone, the standard institutional regimen is permitted.
Drug: Copanlisib (BAY80-6946) — BAY80-6946 (0.6 mg/kg in Cohort 1, 0.8 mg/kg in Cohort 2, 3 and 4) as 60-minute iv infusion once weekly on Days 2, 9, 16 and 23 (Day 23 in Cohort 1, 2 and 3 only) in 28-day cycles

SUMMARY:
This open label Phase 1 study involves treating subjects with advanced cancer with BAY80-6946 in combination with paclitaxel. It will determine the maximum tolerated dose (MTD) and the recommended Phase 2 dose (RP2D) of BAY80-6946 in combination with paclitaxel. The trial will involve multiple participating sites from the US. Following determination of the MTD, an expansion cohort of 20 evaluable subjects with breast cancer was planned. Finally, 16 patients have been enrolled to treatment (Cohort 3). A new expansion cohort with modified dosing cohort is now introduced (Cohort 4: breast cancer expansion cohort with modified dosing) in which another 20 subjects are planned to be enrolled to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have defined tumor classification (ie, TNBC, HER2+ or Luminal) for enrollment. If tumor classification is not available the subject cannot be enrolled. Tumor classification can be based on analysis of archived tumor tissue, or analysis of tumor tissue collected at any time proximal to screening. Subject profile can also be derived from analysis of fresh tumor tissue obtained during screening. Shipment of specimens (archival or fresh tumor tissue, blood, and plasma) to a central lab can take place after subject enrollment.
* No prior paclitaxel treatment for subjects in the dose escalation phase. MTD cohort expansion subjects may have had prior paclitaxel, but must not have experienced moderate or severe hypersensitivity reactions to the drug. Peripheral neuropathy must be Grade ≤ 1.
* Histological or cytological documentation of non-hematologic malignant solid tumor, excluding primary brain or spinal tumors. Patients with prior central nervous system metastases are eligible if all of the following apply: -- Definitive treatment for all lesions (eg, surgery, radiation) was completed at least three months prior to enrollment -- All lesions must be stable or improving on MRI scan performed within one month of enrollment -- All symptoms of the prior CNS metastases are stable.
* At least one measurable lesion or evaluable disease, as per RECIST 1.1
* ECOG Performance Status Assessment of 0 or 1
* Life expectancy of at least 12 weeks

Exclusion Criteria:- History of moderate to severe hypersensitivity (allergy) to drugs formulated in Cremophor® EL (polyoxyethylated castor oil), such as vitamin K, cyclosporin for injection concentrate and teniposide for injection concentrate

* Pre-existing interstitial lung disease and/or severe impaired pulmonary function
* History of cardiac disease; congestive heart failure (CHF) >NYHA Class II; active coronary artery disease, myocardial infarction within 6 months prior to study entry; new onset angina within 3 months prior to study entry or unstable angina, or ventricular cardiac arrhythmias requiring anti-arrhythmic therapy
* Prior diagnosis of Type 1 or 2 diabetes mellitus, hyperglycemia (defined as consistent fasting blood or plasma glucose > 125 mg/dL) or HgBA1c ≥ 7%
* Active clinically serious infections Grade ≥ 2 (NCI-CTCAE version 4.0), including viral hepatitis
* Poorly controlled seizure disorder
* Poorly controlled hypertension, defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management
* Known human immunodeficiency virus (HIV) infection or chronic hepatitis C or B
* Subjects undergoing renal dialysis
* Known bleeding diathesis
* Pregnant or breast feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2011-08-24 (Actual); Primary Completion 2014-10-22 (Actual); Study Completion 2015-06-29 (Actual)

PRIMARY OUTCOMES:
Adverse event collection | Up to 3 years or longer if indicated
Maximum tolerated dose, measured by adverse event profile | Up to 3 years or longer if indicated
Pharmacokinetics characterized by Cmax of BAY80-6946 (and its metabolite(s), if needed) | Multiple time points up to 6 weeks
  Cmax: maximum drug concentration in plasma after single dose administration
Pharmacokinetics characterized by Cmax/D of BAY80-6946 (and its metabolite(s), if needed) | Multiple time points up to 6 weeks
  Cmax/D: Cmax divided by total dose in [mg]
Pharmacokinetics characterized by tmax of BAY80-6946 (and its metabolite(s), if needed) | Multiple time points up to 6 weeks
  tmax: time to reach maximum drug concentration in plasma after single (first) dose
Pharmacokinetics characterized by AUC(0-tlast) of BAY80-6946 (and its metabolite(s), if needed) | Multiple time points up to 6 weeks
  AUC(0-tlast): AUC from time 0 to the last data point above lower limit of quantification
Pharmacokinetics characterized by AUC (if possible) of BAY80-6946 (and its metabolite(s), if needed) | Multiple time points up to 6 weeks
  AUC: area under the plasma concentration vs time curve from zero to infinity
Pharmacokinetics characterized by AUC/D of BAY80-6946 (and its metabolite(s), if needed) | Multiple time points up to 6 weeks
  AUC/D: AUC divided by total dose in [mg]
Pharmacokinetics characterized by half-life of BAY80-6946 (and its metabolite(s), if needed) | Multiple time points up to 6 weeks
Pharmacokinetics characterized by partial AUC values [eg, AUC(0-25)] of BAY80-6946 (and its metabolite(s), if needed) | Multiple time points up to 6 weeks
  AUC(0-25): area under the plasma concentration vs time curve from zero to 25 h p.a.
Pharmacokinetics characterized by clearance of BAY80-6946 (and its metabolite(s), if needed) | Multiple time points up to 6 weeks
Pharmacokinetics characterized by volume of distribution of BAY80-6946 (and its metabolite(s), if needed) | Multiple time points up to 6 weeks
Estimation of percent of dose excreted [unchanged or as metabolites, if relevant) renally during 0 - 25 h after start of BAY80-6946 infusion (AE,ur(0-25)] (for Cohort 4 only) | Multiple time points up to 6 weeks
  AE,ur(0-25): amount of drug excreted via urine during the collection interval 0 - 25 h
Pharmacokinetics characterized by Cmax of Paclitaxel and 6-OH paclitaxel | Multiple time points up to 6 weeks
Pharmacokinetics characterized by tmax of Paclitaxel and 6-OH paclitaxel | Multiple time points up to 6 weeks
Pharmacokinetics characterized by AUC(0-t) of Paclitaxel and 6-OH paclitaxel | Multiple time points up to 6 weeks
Pharmacokinetics characterized by AUC of Paclitaxel and 6-OH paclitaxel | Multiple time points up to 6 weeks
Pharmacokinetics characterized by half-life of Paclitaxel and 6-OH paclitaxel | Multiple time points up to 6 weeks
Pharmacokinetics characterized by clearance of Paclitaxel and 6-OH paclitaxel | Multiple time points up to 6 weeks
Pharmacokinetics characterized by volume of distribution (If possible and needed) of Paclitaxel and 6-OH paclitaxel | Multiple time points up to 6 weeks
Effect of BAY80-6946 on paclitaxel PK will be assessed by comparing Cmax of Cycle 1 Day 1 and Cycle 1 Day 15 | Multiple time points up to 6 weeks
Effect of BAY80-6946 on paclitaxel PK will be assessed by comparing AUC(0-tlast) of Cycle 1 Day 1 and Cycle 1 Day 15 | Multiple time points up to 6 weeks

SECONDARY OUTCOMES:
Number of patients with mutational status | Up to 3 years or longer if indicated
Tumor Response as measured by RECIST 1.1 criteria | Up to 3 years or longer if indicated

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- United States (3):
  - St Louis, Missouri
  - New York, New York
  - Houston, Texas